CLINICAL TRIAL: NCT01092832
Title: A Prospective, Open-label, Non-comparative Study To Assess The Safety, Tolerability And Efficacy Of Voriconazole For The Primary And Salvage Treatment Of Invasive Candidiasis, Candidemia, And Esophageal Candidiasis In Pediatric Subjects
Brief Title: A Study Of The Safety, Tolerability And Effective Of Voriconazole For The Treatment Of Serious Candida Infection And Candida Infection Of The Throat In Pediatric Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This protocol terminated prematurely on July 8, 2013 due to slow enrollment, not because of any safety issues or concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A1501085; 2009-012848-16 (EudraCT Number)
Record Dates: First submitted 2010-03-10; First posted 2010-03-25 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Candidiasis
Keywords: Invasive Candidiasis Candidemia Esophageal Candidiasis
MeSH Terms: conditions — Candidiasis | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active voriconazole (Experimental): All subjects in this study will receive active voriconazole in an open-label fashion; there is no comparator in this study.
  Interventions: Drug: voriconazole

INTERVENTIONS:
Drug: voriconazole — Subjects 12 - <18 yrs (excluding subjects 12 - 14 yrs weighing <50kg): For IC, the loading dose is 6 mg/kg IV q12h on Day 1, followed by 4 mg/kg IV q12h thereafter. Oral therapy, if given, will be administered at a dose of 200 mg q12h. For EC, no loading dose is required, and subjects will be initiated on 3 mg/kg IV q12h. Oral therapy, if given, will be administered at a dose of 200 mg q12h.
  Subjects 2 - <12 yrs, and subjects 12 - 14 weighing <50kg: For IC, the loading dose is 9 mg/kg IV q12h on Day 1, followed by 8 mg/kg IV q12h thereafter. For EC, no loading dose is required, and subjects will be initiated on 4 mg/kg IV q12. Oral therapy, if given, will be administered at a dose of 9 mg/kg q12h (maximum initial dose of 300 mg).
  Subjects will be treated for a minimum of 14 days for invasive candidiasis/candidemia or a minimum of 7 days for esophageal candidiasis. Subjects will be treated for up to a maximum of 42 days.
  Other Names: Vfend

SUMMARY:
The purpose of this study is to determine whether voriconazole is safe and effective for the treatment of serious Candida infection and Candida infection of the esophagus in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 2 to <18 years of age; Subjects 2 to <12 years of age will be permitted to enroll in this study only after a Pfizer sponsored pharmacokinetic study confirms the proposed dosage corresponding to this age group is appropriate.
* Patients with confirmed Candida infection of the blood, body tissues, or the esophagus.
* Patient's doctor feels voriconazole is an appropriate choice of therapy.

Exclusion Criteria:

* A known allergy to voriconazole or to azole to antifungal drugs.
* Females who are pregnant, lactating (breast feeding) or planning a pregnancy during the course of the study, or who are of childbearing potential and not using highly effective method of birth control.
* A patient who is receiving treatment with a drug know to interfere with the heart's electrical system (QTc prolongation).
* A patient who is receiving treatment with a drug that is not permitted to be used with voriconazole.
* For primary therapy: a patient who has received more than 48 hours of antifungal therapy for the current episode of Candida infection.
* A patient with significant underlying liver disease at the time of enrollment in the study.
* A patient with significant renal disease (CrCl < 50 ml/min) at the time of enrollment in the study.
* A patient with a high likelihood of death within 72 hours of study enrollment due to factors unrelated to Candida infection.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- China (2):
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Beijing Children's Hospital, Capital University of Medical Sciences, Beijing
- Fakultni nemocnice Brno - Klinika detske onkologie, Brno, Czechia
- Hong Kong (3):
  - Department of Paediatrics and Adolescent Medicine, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin, N.T.
- Hungary (3):
  - Semmelweis Egyetem, II. sz. Szemeszeti Klinika, Budapest
  - Semmelweis Egyetem, II. sz. Gyermekgyogyaszati Klinika, Budapest
  - Fovarosi Onkormanyzat Egyesitett Szent Istvan és Szent Laszlo Korhaz-Rendelointezet, Budapest
- Instituto Nacional de Pediatria, Colonia Insurgentes Cuicuilco, Delegacion Coyoacan, Mexico City, Mexico
- Philippines (2):
  - Medical Research Laboratory Philippine General Hospital University of the Philippines, Ermita, Manila
  - Rm. 112 ICHHD, National Institutes of Health-University of the Philippines Manila, Manila
- Oddzial Pediatryczny I- Hematologiczno-Onkologiczny, Olsztyn, Poland
- Detska fakultna nemocnica s poliklinikou Bratislava, Bratislava, Slovakia

REFERENCES:
- [Derived] Martin JM, Macias-Parra M, Mudry P, Conte U, Yan JL, Liu P, Capparella MR, Aram JA. Safety, Efficacy, and Exposure-Response of Voriconazole in Pediatric Patients With Invasive Aspergillosis, Invasive Candidiasis or Esophageal Candidiasis. Pediatr Infect Dis J. 2017 Jan;36(1):e1-e13. doi: 10.1097/INF.0000000000001339. PMID 27636722
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501085&StudyName=A%20Study%20Of%20The%20Safety%2C%20Tolerability%20And%20Effective%20Of%20Voriconazole%20For%20The%20Treatment%20Of%20Serious%20Candida%20Infection%20And%20Candida%20Infection

RESULTS

PARTICIPANT FLOW:
Groups:
- Voriconazole: 2 to <12 Years: Participants aged 2 to less than (<)12 years (and young adolescents aged 12 to 14 years weighing <50 kilograms [kg]) with invasive candidiasis/candidemia (ICC) received a loading dose of voriconazole 9 milligrams per kg (mg/kg), intravenously (IV), every 12 hours (q12h) for the first 24 hours, followed by maintenance dosing of voriconazole 8 mg/kg, IV, q12h for a minimum of 5 days of IV therapy. Participants with esophageal candidiasis (EC) received voriconazole 4 mg/kg, IV, q12h for a minimum of 5 days of IV therapy. In both ICC and EC, once signs and symptoms of Candida infection had resolved and the participant was clinically stable, participants were switched to oral (PO) therapy and received voriconazole 9 mg/kg, PO, q12h (maximum dose of 350 mg). Voriconazole was administered for at least 7 days (participants with EC) or 14 days (participants with ICC) after last positive blood culture up to a maximum of 42 days of treatment.
- Voriconazole: 12 to <18 Years: Participants aged 12 to <18 years (excluding those aged 12-14 years weighing <50 kg) with ICC received a loading dose of voriconazole 6 mg/kg, IV, q12h for the first 24 hours, followed by maintenance dosing of voriconazole 4 mg/kg, IV, q12h for a minimum of 7 days of IV therapy. Participants with EC received voriconazole 3 mg/kg, IV, q12h for a minimum of 5 days of IV therapy. In both ICC and EC, once signs and symptoms of Candida infection had resolved and the participant was clinically stable, participants were switched to PO therapy and received voriconazole 200 mg, PO, q12h. Voriconazole was administered for at least 7 days (participants with EC) or 14 days (participants with ICC) after last positive blood culture up to a maximum of 42 days of treatment.
Period: Overall Study
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Started | 14 | 8
Completed | 13 | 8
Not Completed | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of study medication.
Groups:
- Voriconazole: 2 to <12 Years: Participants aged 2 to <12 years (and young adolescents aged 12 to 14 years weighing <50 kg) with ICC received a loading dose of voriconazole 9 mg/kg), IV, q12h for the first 24 hours, followed by maintenance dosing of voriconazole 8 mg/kg, IV, q12h for a minimum of 5 days of IV therapy. Participants with EC received voriconazole 4 mg/kg, IV, q12h for a minimum of 5 days of IV therapy. In both ICC and EC, once signs and symptoms of Candida infection had resolved and the participant was clinically stable, participants were switched to PO therapy and received voriconazole 9 mg/kg, PO, q12h (maximum dose of 350 mg). Voriconazole was administered for at least 7 days (participants with EC) or 14 days (participants with ICC) after last positive blood culture up to a maximum of 42 days of treatment.
- Total: Total of all reporting groups
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years | Total
Number analyzed (Participants) | 14 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.8 (2.9) | 14.4 (1.7) | 9.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events - Overall Summary
Description: Percentage of participants with adverse events (AEs), serious adverse events (SAEs), severe AEs, who discontinued due to AEs, or who had dose redued or temporarily discontinued due to AEs.
Time Frame: Baseline up to 1 month follow-up
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Number analyzed (Participants) | 14 | 8
percentage of participants
  With AEs | 92.9 | 75.0
  With SAEs | 14.3 | 12.5
  With severe AEs | 28.6 | 37.5
  Discontinued due to AEs | 14.3 | 25.0
  Dose reduced/temporary discontinuation due to AE | 21.4 | 0

2. Secondary Outcome: Percentage of Participants With a Global Response of Success at End of Treatment (EOT)
Description: Global response was determined programmatically based on investigator assessment of clinical and microbiological response. Global response of success was defined as clinical cure or improvement AND microbiological eradication or presumed eradication. Exact 95 percent (%) confidence interval for binomial proportions using Clopper-Pearson method.
Time Frame: EOT (from 7 to 42 days of treatment)
Population: Modified Intent-to-Treat (MITT) Population: all participants who received at least 1 dose of study medication and who have confirmed ICC, EC or participants with EC who do not have confirmation of EC by esophagoscopy, but who had at least confirmation of oropharyngeal candidiasis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Number analyzed (Participants) | 9 | 8
percentage of participants | 88.9 [51.75 to 99.72] | 62.5 [24.49 to 91.48]

3. Secondary Outcome: All-Cause Mortality - Number of Participant Deaths
Time Frame: Day 28 and 1 Month Follow-up
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Number analyzed (Participants) | 14 | 8
participants
  Day 28 | 0 | 0
  1 Month Follow-up | 0 | 0

4. Secondary Outcome: Time to Death
Time Frame: Baseline up to 1 month follow-up
Population: No participants died within the safety reporting period, therefore time to death was not applicable.
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 49 (7 days after the last dose of study drug)
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Voriconazole: 2 to <12 Years | Voriconazole: 12 to <18 Years
Serious Adverse Events (participants affected / at risk) | 2/14 | 1/8
Other Adverse Events (participants affected / at risk) | 13/14 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole: 2 to <12 Years (N=14) | Voriconazole: 12 to <18 Years (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Splenic candidiasis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole: 2 to <12 Years (N=14) | Voriconazole: 12 to <18 Years (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypothrombinaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Platelet disorder (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Amaurosis (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Corneal opacity (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Eyelid disorder (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 2 | 1
Retinal disorder (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Device occlusion (General disorders) | 0 | 1
Hypothermia (General disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 1
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Anorectal cellulitis (Infections and infestations) | 1 | 0
Bone abscess (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Splenic candidiasis (Infections and infestations) | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase abnormal (Investigations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase abnormal (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phophatase abnormal (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1
Drug level decreased (Investigations) | 0 | 1
Gamma-glutamyltransferase abnormal (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Haematocrit abnormal (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Lymphocyte percentage abnormal (Investigations) | 1 | 0
Monocyte count abnormal (Investigations) | 1 | 0
Staphylococcus test positive (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Testicular mass (Reproductive system and breast disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Phlebitis (Vascular disorders) | 0 | 1
Venoocclusive disease (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to slow enrollment. The study was not terminated due to any safety issues or concerns. Interpretation of the data are limited due to the small sample size and descriptive design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. PI will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. PI may not disclose previously undisclosed confidential information other than study results.